CLINICAL TRIAL: NCT03637712
Title: Deep-Learning for Automatic Polyp Detection During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-00746
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Screening Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening Colonoscopy (Experimental): Patients undergoing standard screening or surveillance colonoscopy will be included
  Interventions: Device: Computer Algorithm

INTERVENTIONS:
Device: Computer Algorithm — This device is a computer algorithm that runs in the background during routine screening or surveillance colonoscopy that is designed to aid in the detection of polyps

SUMMARY:
The primary objective of this study is to examine the role of machine learning and computer aided diagnostics in automatic polyp detection and to determine whether a combination of colonoscopy and an automatic polyp detection software is a feasible way to increase adenoma detection rate compared to standard colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for routine colonoscopy for screening and/or surveillance purposes.
* Ability to provide written, informed consent and understand the responsibilities of trial participation

Exclusion Criteria:

* People with diminished cognitive capacity.
* The subject is pregnant or planning a pregnancy during the study period.
* Patients undergoing diagnostic colonoscopy (e.g. as an evaluation for active GI bleed)
* Patients with incomplete colonoscopies (those where endoscopists did not successfully intubate the cecum due to technical difficulties or poor bowel preparation)
* Patients that have standard contraindications to colonoscopy in general (e.g. documented acute diverticulitis, fulminant colitis and known or suspected perforation).
* Patients with inflammatory bowel disease
* Patients with any polypoid/ulcerated lesion > 20mm concerning for invasive cancer on endoscopy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate | 1 Day
  the proportion of colonoscopic examinations performed that detect one or more polyp

CONTACTS AND LOCATIONS:
Overall Officials: Seth Gross, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States